CLINICAL TRIAL: NCT02280304
Title: Neuroimaging Meditation Therapy in Veterans With Co-Morbid TBI and PTSD
Brief Title: Meditation in Veterans With PTSD and Mild TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Palo Alto University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D1608-P; I21RX001608-01A1 (NIH)
Record Dates: First submitted 2014-10-17; First posted 2014-10-31 (Estimated); Results first posted 2020-03-09 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-02

CONDITIONS: Stress Disorders, Post-Traumatic; Concussion, Mild
Keywords: Stress Disorders, Post-Traumatic; Concussion, Mild; Brain Injuries; Community Integration; Meditation; Magnetic Resonance Imaging
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Brain Concussion; Brain Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inner Resources for Veterans (IRV) mindfulness and mantra (Experimental): Complete a mindfulness and mantra therapy
  Interventions: Behavioral: Inner Resources for Veterans (IRV)
- Essential Skills therapy (Active Comparator): Learn symptoms of mTBI and PTSD, coping skills
  Interventions: Behavioral: Essential Skills therapy

INTERVENTIONS:
Behavioral: Inner Resources for Veterans (IRV) — Mindfulness and breath-focused mantra therapy which uses techniques that encourage present moment attention for the purpose of improving self-monitoring and self-regulation
  Arms: Inner Resources for Veterans (IRV) mindfulness and mantra
Behavioral: Essential Skills therapy — This active comparator is adapted from a therapy utilized at multiple VAs as a psychoeducational AND symptom management treatment for PTSD. In it, participants learn about mTBI and PTSD symptoms and coping information for PTSD.
  Arms: Essential Skills therapy

SUMMARY:
The goal of this study is to learn more about how Inner Resources for Veterans (IRV), a mindfulness and mantra therapy, helps Veterans with Post Traumatic Stress Disorder (PTSD) and mild traumatic brain injury (mTBI). PTSD is a disorder that occurs after exposure to one or more emotionally traumatic experiences. People with PTSD may experience anxiety, pay extra attention to their surroundings, involuntarily remember their traumatic experiences, and/or want to avoid situations where these symptoms are increased. MTBI may result from being in a blast explosion, with pressure from the blast potentially disrupting the brain's structure and function. At this time, it is not well known how PTSD and mTBI may affect each other.

In this study, the investigators will be looking at the behavioral and neurological changes (changes in the brain) and the reductions in PTSD symptoms that may come from participating in this treatment. The investigators are interested in determining if treatment does reverse changes in the brain caused by PTSD and mTBI. To help the investigators understand changes in how the brain functions, the participants will complete a functional magnetic resonance imaging (fMRI) scan before and after either IRV or an active control group. Both conditions are 9-session, 12-week interventions. Participation will help the investigators understand how therapy for PTSD and mTBI impacts the brain's response to emotions and therapeutic processes.

DETAILED DESCRIPTION:
Approximately 18-22% of Operation Enduring Freedom/Operation Iraqi Freedom/ Operation New Dawn (OEF/OIF/OND) Veterans have been diagnosed with posttraumatic stress disorder (PTSD), and 15-30% of Veterans report mild traumatic brain injury (mTBI). The effects of mTBI and PTSD have been evident since military personnel first came home and continue to be difficult to eradicate. At 3-4 months post-deployment, OIF Veterans with mild TBI were more likely to endorse PTSD symptoms than those without mTBI. The co-morbidity may be long-lasting, or at least recurrent, as TBI-related symptoms were strongly associated with traumatic stress five years after injury. In an examination of factors associated with postconcussive symptoms, PTSD was a strong factor. In active duty marines, mTBI during deployment predicted PTSD after deployment, and in a study of OEF-OIF-OND Veterans, 57.3% of those with mTBI had PTSD.

The literature on how mTBI and co-morbid PTSD affect each other and the effects on Veterans several years post-deployment is sparse. Treatment recommendations specific to Veterans with both mTBI and PTSD are in flux, and while treatments address each disorder independently, they may not be effective when the two disorders co-occur. Further impacting successful treatment of Veterans is the fact that many Veterans do not seek treatment, in part due to the distance they travel to obtain VA services and stigma.

Treatments that are accessible and improve symptoms in patients with mTBI and PTSD alone may facilitate rehabilitation in Veterans with co-morbid mTBI and PTSD. Mindfulness and mantra have been suggested to be effective in Veterans with PTSD and in civilians with TBI, improving quality of life. The current study proposes a type of mindfulness targeted for Veterans, Inner Resources for Veterans (IRV).

Inner Resources for Veterans (IRV), a mindfulness and mantra intervention, is based on Inner Resources for Stress, an intervention which utilizes mindfulness, techniques that encourage present moment attention for the purpose of promoting better self-monitoring and self-regulation, and mantra, the repetition of sounds that do not have meaning in order to maintain present focused attention. The Inner Resources protocol targets PTSD and has been associated with reduced PTSD and anxiety symptoms, reduced number of depressive symptoms, and depression remissions at a 9-month follow-up, as well as increased perceived self-efficacy. Pilot results of older combat Veterans with PTSD indicated that Inner Resources is a safe, feasible, and acceptable intervention. The control condition is an active treatment called Essential Skills, a manualized therapy adapted from a similar therapy utilized at multiple VAs as a psychoeducational and symptom management treatment for PTSD. In a previous study at the Michael E. DeBakey VA that did not investigate the effect of mTBI, Essential Skills provided education on the symptoms and effects of PTSD. For example, subjects learned to recognize the circumstances that triggered their symptoms, how to identify and participate in healthy activities, and how to monitor their sleep. In the current study, in Essential Skills, Veterans learn about symptoms of both mTBI and PTSD and coping skills.

In addition to the changes in functional and psychological symptoms and neural pathways, IRV would offer Veterans a treatment they could utilize whenever challenging situations occur regardless of location. Since the treatment would be relatively cost-free after initial training, IRV could also dramatically reduce financial burden to both Veterans and VA. Few treatment studies focusing on Veterans with co-morbid mTBI and PTSD support the innovation of this study, as does generation of community integration data to relate to changes in functional connectivity.

ELIGIBILITY:
Inclusion Criteria:

* Mild traumatic brain injury (mTBI) as defined by the VA/DoD Clinical Practice Guideline.
* PTSD as assessed by the Clinician Administered PTSD Scale (CAPS);
* Aged 18 - 49;
* Have not previously participated in meditation training.

Exclusion Criteria:

The investigators will exclude subjects who:

* Meet DSM-IV criteria for drug or alcohol abuse in past 30 days;
* Have a history of severe TBI based on any of following:

  * Glasgow Coma Score < 8;
  * alteration of consciousness greater than 24 hours; loss of consciousness greater than 30 minutes;
* Have current neurological or general medical conditions known to impact cognitive and/or emotional functioning, including but not limited to:

  * epilepsy,
  * Parkinson's disease,
  * Huntington's disease,
  * Alzheimer's disease,
  * stroke,
  * chemotherapy for cancer;
* Have acute psychological instability as assessed by MEDVAMC clinician or study staff or concurrent diagnosis or schizophrenia, schizoaffective disorder, delusional disorder, organic psychosis, and subjects taking antipsychotic medication, and
* Have already completed a course of meditation training.
* The investigators will also exclude participants with general contraindications for MRI, including metal in or around the head (e.g., orthodontia, non-removable body piercings, etc.), ferromagnetic material in the body (e.g., non-removable body piercings), or non-MRI compatible medical devices.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2014-11-03 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2018-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary R Newsome, PhD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 364 Veterans were pre-screened. Flyers were posted at the VA and at the University of Houston; however, most of the people who responded had been contacted in Mental Health and Neurology clinics.
Pre-assignment Details: Of 364 Veterans pre-screened, 85 were invited to come in for further eligibility assessment for PTSD, mTBI, and exclusionary disorders. Of these, 33 did not attend or excluded themselves, leaving 46 enrolled. Of these, 9 dropped out before group assignment, and 15 dropped out post group assignment, leaving a total of 22 finishing the study.
Groups:
- Inner Resources for Veterans Meditation Therapy: Participants will complete meditation therapy
  Inner Resources for Veterans (IRV): Meditation therapy which utilizes mindfulness, techniques that encourage non-judgmental attention to oneself in the present moment
- PTSD and mTBI Education: Participants will learn about symptoms and triggers of PTSD and mTBI
  PTSD and mTBI education: Participants will learn about symptoms and triggers of PTSD and mTBI
Period: Overall Study
Arm/Group | Inner Resources for Veterans Meditation Therapy | PTSD and mTBI Education
Started | 19 | 18
Completed | 12 | 10 (A non completer received the allocated intervention before being lost to follow-up.)
Not Completed | 7 | 8
Not completed — Lost to Follow-up | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Inner Resources for Veterans Meditation and Mantra Therapy: Participants complete meditation and mantra therapy
  Inner Resources for Veterans (IRV): Meditation therapy which utilizes mindfulness, techniques that encourage non-judgmental attention to oneself in the present moment
- Essential Skills Therapy: Participants learn about symptoms of PTSD and mTBI and coping skills for PTSD.
- Total: Total of all reporting groups
Arm/Group | Inner Resources for Veterans Meditation and Mantra Therapy | Essential Skills Therapy | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 18 | 37
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (7.2) | 36.1 (5.3) | 36.2 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 5
  Male | 14 | 18 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic | 2 | 5 | 7
  Ethnicity: Not Hispanic | 17 | 13 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: African American | 5 | 8 | 13
  Race: Caucasian | 13 | 9 | 22
  Race: African American and Other | 0 | 1 | 1
  Race: Other | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 18 | 37
PTSD Checklist (PCL5) [Mean (Standard Deviation); unit: units on a scale] — Population: Missing Data. Scores fall in the range 0-80; higher scores indicate worse outcome
  units on a scale
    number analyzed (Participants) | 16 | 12 | 28
    (all) | 47.9 (11.7) | 52.6 (12.3) | 49.8 (12.0)
PHQ-9 Depression [Mean (Standard Deviation); unit: units on a scale] — Population: Missing data. Scores fall in the range 0-27; higher scores indicate worse outcome
  units on a scale
    number analyzed (Participants) | 16 | 12 | 28
    (all) | 15.8 (5.1) | 17.4 (6.4) | 16.5 (5.6)

OUTCOME MEASURES:

1. Primary Outcome: Clinician-Administered PTSD Scale (CAPS5)
Description: Changes in responses in the CAPS5 will be measured in patients following IRV meditation+mantra or ES education control.
Time Frame: 12 weeks
Population: One CAPS rater did not meet study criteria for expert CAPS administration; as a result, the CAPS data are not considered valid.
Groups:
- Inner Resources for Veterans (IRV) Mindfulness and Mantra: Participants will complete meditation and mantra therapy
  Inner Resources for Veterans (IRV): Meditation therapy which utilizes mindfulness, techniques that encourage non-judgmental attention to oneself in the present moment
- Essential Skills Therapy: Participants will learn about symptoms of PTSD and mTBI and coping skills for PTSD
  PTSD and mTBI education: Participants will learn about symptoms and triggers of PTSD and mTBI
Arm/Group | Inner Resources for Veterans (IRV) Mindfulness and Mantra | Essential Skills Therapy
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Participants With Significant Changes in Resting State Functional Connectivity Following Meditation or Control
Description: Functional connectivity was measured between the Default Mode Network (DMN) and lateral prefrontal cortex (LPFC), and between the amygdala and anterior cingulate. There were four seeds for the DMN (MPFC, PCC, left lateral parietal, right lateral parietal), and two seeds for the amygdala (right and left). Correlation coefficients representing the degree of connectivity between hypothesized regions were Fisher transformed. An a priori threshold of p<.001 at the voxel level and p<.05, FDR corrected for multiple comparisons across the whole brain, at the cluster level were used to determine significant connectivity.
Time Frame: 12 weeks and baseline
Population: The sample sizes here differ from those reported for other measures because these are the numbers of subjects who had MRI available and with acceptable quality assessment (i.e., not excluded because of excessive motion or sleepiness) for both time periods.
Measure: Count of Participants; unit: Participants
Groups:
- Inner Resources for Veterans (IRV) Mindfulness and Mantra: Participants will complete meditation therapy
  Inner Resources for Veterans (IRV): Meditation therapy which utilizes mindfulness, techniques that encourage non-judgmental attention to oneself in the present moment
Arm/Group | Inner Resources for Veterans (IRV) Mindfulness and Mantra | Essential Skills Therapy
Number analyzed (Participants) | 9 | 11
Participants
  DMN (MPFC seed) to LPFC | 0 | 0
  DMN (PCC seed) to LPFC | 0 | 0
  DMN (RLP seed) to LPFC | 0 | 0
  DMN (LLP seed) to LPFC | 0 | 0
  Amygdala (right) to ACC | 0 | 0
  Amygdala (left) to ACC | 0 | 0
Statistical Analysis 1: Comparison: Inner Resources for Veterans (IRV) Mindfulness and Mantra vs Essential Skills Therapy; Z-scores represent Fisher transformed correlation coefficients representing the correlations between hypothesized regions. Positive values represents positive connectivity between regions. Negative values represent anticorrelations, or negative relations, between hypothesized regions; Test type: Superiority; p > 0.05, t-test, 1 sided — A priori threshold = voxel p<.001, cluster p<.05, FDR whole brain correction. There is no correction for multiple seeds given small sample sizes and pre-post design. To report NS p-values and associated z-scores, uncorrected cluster ps were queried

3. Secondary Outcome: Community Reintegration in Service Members (CRIS)
Description: Scores at baseline and 12 weeks in responses to the computerized version of the Community Reintegration in Service Members (CRIS-CAT) questionnaire in patients following meditation or control. There are three subscales: Extent of Participation (range 24-90), Perceived Limitations (range 33-99), and Satisfaction (range 34-91). Higher is better.
Time Frame: 12 weeks and baseline
Population: The sample sizes here differ from those reported for other measures because these are the numbers of subjects who had completed the CRIS at both time periods.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Essential Skills Therapy | Inner Resources for Veterans (IRV) Mindfulness and Mantra
Number analyzed (Participants) | 8 | 8
score on a scale
  Baseline Extent of Participation | 34.1 (5.3) | 36.4 (3.7)
  Baseline Perceived Limitations | 37.3 (3.5) | 38.9 (4.6)
  Baseline Satisfaction | 38.0 (3.9) | 38.4 (3.4)
  12 weeks Extent of Participation | 34.9 (6.0) | 38.2 (6.2)
  12 weeks Perceived Limitations | 39.1 (3.5) | 39.7 (3.3)
  12 weeks Satisfaction | 38.6 (5.1) | 39.7 (5.3)
Statistical Analysis 1: Comparison: Inner Resources for Veterans (IRV) Mindfulness and Mantra; Test type: Other; Mean Difference (Net) = 1.8
Statistical Analysis 2: Comparison: Inner Resources for Veterans (IRV) Mindfulness and Mantra; Test type: Other; Cohen's d = 0.35 — Cohen's d reflects Extent of Participation subscale of the CRIS, Post - Pre
Statistical Analysis 3: Comparison: Essential Skills Therapy; Test type: Other; Median Difference (Net) = .8
Statistical Analysis 4: Comparison: Essential Skills Therapy; Test type: Other; Cohen's d = .14 — Cohen's d reflects Extent of Participation Scale of the Cris pre- post
Statistical Analysis 5: Comparison: Inner Resources for Veterans (IRV) Mindfulness and Mantra; Test type: Other; Median Difference (Net) = .8
Statistical Analysis 6: Comparison: Inner Resources for Veterans (IRV) Mindfulness and Mantra; Test type: Other; Cohen's d = .20 — Cohens d reflects the Cris pre post Perceived Limitations scale
Statistical Analysis 7: Comparison: Essential Skills Therapy; Test type: Other; Mean Difference (Net) = 1.8
Statistical Analysis 8: Comparison: Essential Skills Therapy; Test type: Other; Cohens d = .53
Statistical Analysis 9: Comparison: Inner Resources for Veterans (IRV) Mindfulness and Mantra; Test type: Other; Mean Difference (Net) = 1.3
Statistical Analysis 10: Comparison: Inner Resources for Veterans (IRV) Mindfulness and Mantra; Test type: Other; Cohens d = .29
Statistical Analysis 11: Comparison: Essential Skills Therapy; Test type: Other; Mean Difference (Net) = .6
Statistical Analysis 12: Comparison: Essential Skills Therapy; Test type: Other; Cohens d = .13

4. Other Pre Specified Outcome: PTSD Checklist 5 (PCL5) Difference Score
Description: The PTSD Checklist 5 (PCL5) is a measure of PTSD symptoms based on DSM-V. The scores fall in the range 0-80; higher scores indicate worse outcome. We calculated the PTSD Checklist 5 (PCL5) difference score by subtracting the value at baseline minus the value at week 12. In this case higher scores represent a reduction in PTSD symptoms.
Time Frame: 12 weeks, baseline
Population: The sample sizes here differ from those reported for other measures because these are the numbers of subjects who had completed PCL-5 at both time periods.
Measure: Mean (Full Range); unit: Score on a scale
Groups:
- Essential Skills Therapy: Participants will learn about symptoms of PTSD and mTBI and coping skills for PTSD.
Arm/Group | Inner Resources for Veterans (IRV) Mindfulness and Mantra | Essential Skills Therapy
Number analyzed (Participants) | 10 | 7
Score on a scale | 11.77 [0 to 80] | 5.58 [0 to 80]
Statistical Analysis 1: Comparison: Inner Resources for Veterans (IRV) Mindfulness and Mantra vs Essential Skills Therapy; Cohen's d effect sizes are reported for changes over time (0 weeks vs. 12 weeks) in each group separately; Test type: Other; Cohens d = .86 — Cohen's d effect size (Cohen's d=.20 small, Cohen's d=.50 medium, Cohen's d=.80 large)
Statistical Analysis 2: Comparison: Essential Skills Therapy; Cohen's d effect sizes are reported for changes over time (0 weeks vs. 12 weeks) in each group separately; Test type: Other; Cohens d = .30 — Cohen's d effect size (Cohen's d=.20 small, Cohen's d=.50 medium, Cohen's d=.80 large)

5. Other Pre Specified Outcome: Patient Health Questionnaire-9 (PHQ-9) Patient Depression Questionnaire Difference Score
Description: The Patient Health Questionnaire-9 (PHQ-9) measure is a self-report measure of depression symptoms. Scores fall in the range 0-27; higher scores indicate worse outcome. This difference score denotes improvement in symptoms of depression. It was calculated by subtracting the value of PHQ-9 scores at baseline minus PHQ-9 scores scores at week 12.
Time Frame: 12 weeks, baseline
Population: The sample sizes here differ from those reported for other measures because these are the numbers of subjects who had PHQ-9 forms completed at both time periods.
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Inner Resources for Veterans (IRV) Mindfulness and Mantra | Essential Skills Therapy
Number analyzed (Participants) | 10 | 7
Score on a scale | 5.0 [0 to 27] | 2.0 [0 to 27]
Statistical Analysis 1: Comparison: Inner Resources for Veterans (IRV) Mindfulness and Mantra vs Essential Skills Therapy; Cohen's d effect sizes are reported for changes over time (0 weeks vs. 12 weeks) in each group separately; Test type: Other; Cohens d = 1.32 — Cohen's d effect size change (Cohen's d =0.20 is a small effect; Cohen's d=0.50 is a medium effect; Cohen's d=0.80 is a large effect.)
Statistical Analysis 2: Comparison: Essential Skills Therapy; Cohen's d effect sizes are reported for changes over time (0 weeks vs. 12 weeks) in each group separately; Test type: Other; Cohens d = .27 — Cohen's d effect size (Cohen's d =0.20 is a small effect; Cohen's d=0.50 is a medium effect; Cohen's d=0.80 is a large effect.)

6. Post Hoc Outcome: Test of Additional Limbic Seeds (Hippocampal and Parahippocampal Gyri)
Description: Within-group Post vs. Pre t-tests were done for each group with left and right hippocampal and parahippocampal gyrus (PHG) as seeds. Below are mean Fisher-transformed z scores and respective standard deviations of the Pearson's product correlation coefficients between the seed and cluster for each group. Positive mean z-scores scores reflect positive correlations between the seed and the cluster, and negative mean z-scores reflect negative correlations between the seed and the cluster. L IPL = left intraparietal lobule; VMPFC=ventromedial prefrontal cortex
Time Frame: 12 weeks
Population: The sample sizes here differ from those reported for other measures because these are the numbers of subjects who had MRI available and with acceptable quality assessment (i.e., not excluded because of excessive motion or sleepiness) for both time periods. Note that the sample sizes are identical to those reported in the secondary outcome section.
Measure: Mean (Standard Deviation); unit: z-scores
Groups:
- Inner Resources for Veterans (IRV) Mindfulness and Mantra: Meditation and mantra therapy
- Essential Skills Therapy: Control therapy involving learning about PTSD and mTBI symptoms and coping information.
Arm/Group | Inner Resources for Veterans (IRV) Mindfulness and Mantra | Essential Skills Therapy
Number analyzed (Participants) | 11 | 9
z-scores | 0.17 (0.07) | 0.15 (0.03)
Statistical Analysis 1: Comparison: Inner Resources for Veterans (IRV) Mindfulness and Mantra; Test type: Superiority; p < .0099, t-test, 2 sided — The p-value obtained for the L PHG seed/L IPL cluster is 0.0099. The critical p-value after Bonferroni correction for multiple seeds is p=.008; Significance is determined when clusters reach voxel threshold p<.001, cluster p<.05 FDR corrected for multiple comparisons across the whole brain
Statistical Analysis 2: Comparison: Essential Skills Therapy; Test type: Superiority; p < 0.02, t-test, 2 sided — The p-value obtained for the L anterior PGH seed/left VMPC cluster is 0.02. The critical p-value after Bonferroni correction for six seeds is p=.008; [statistical method as in outcome 6, analysis 1]

7. Post Hoc Outcome: Relating Extent of Participation in the Community (as Measured by the CRIS-CAT) Prior to Therapy to the Functional Connectivity of the Right Hippocampus After Therapy.
Description: The goal was to see if extent of participation in the community prior to therapy could predict the degree of functional connectivity between regions whose connectivity has been suggested to be part of a context processing network, disrupted during PTSD. The hippocampus was investigated because it is one of these regions. (The MPFC and thalamus are others.)
Time Frame: 12 weeks
Population: Groups were combined to increase range of the sample size and to examine the general effect of therapy. Subjects (n=16; 9 IRV and 7 ES) were those who had both a post-therapy scan (regardless of therapy, IRV or ES) and CRIS-CAT scores prior to therapy.
Measure: Number; unit: beta
Groups:
- Combined Groups (IRV + ES): Groups were combined to increase range of the sample size and to examine the general effect of therapy. Subjects (n=16; 9 IRV and 7 ES) were those who had both a post-therapy scan (regardless of therapy, IRV or ES) and CRIS-CAT scores prior to therapy. Analysis: Pre-therapy scores were regressed onto post-therapy functional connectivity, relative to pre-therapy functional connectivity (Post-Pre).
Arm/Group | Combined Groups (IRV + ES)
Number analyzed (Participants) | 16
beta | 0.02
Statistical Analysis 1: Comparison: Combined Groups (IRV + ES); The extent of community participation prior to therapy was correlated with the functional connectivity of the right hippocampus seed after therapy (post-pre); Test type: Other; p < .000038, Regression, Linear — Cluster in MPFC p<0.000038 FDR corrected for multiple comparisons across whole brain. Bonferroni correction for multiple seeds p=0.008; Significance is determined when voxel (height) threshold p=.001, cluster threshold p=.05, FDR corrected for multiple tests across the whole brain; Slope = 0.02
Statistical Analysis 2: Comparison: Combined Groups (IRV + ES); [analysis description as in outcome 7, analysis 1]; Test type: Other; p < 0.000149, Regression, Linear — Cluster in the right cerebellum (crus 2) p<0.000149 FDR corrected for multiple comparisons across the whole brain. Bonferroni for multiple seeds p=0.008; [statistical method as in outcome 7, analysis 1]; Slope = 0.02

ADVERSE EVENTS:
Time Frame: 39 MONTHS
Arm/Group | Inner Resources for Veterans Meditation Therapy | PTSD and mTBI Education
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 0/19 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2016-10-04): https://cdn.clinicaltrials.gov/large-docs/04/NCT02280304/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-03-02): https://cdn.clinicaltrials.gov/large-docs/04/NCT02280304/Prot_SAP_001.pdf